CLINICAL TRIAL: NCT06264960
Title: The Effect of Music Therapy and Breathing Exercise on Anxiety and Pain in Patients Undergoing Coronary Angiography: A Randomised Controlled Study
Brief Title: The Effect of Music Therapy and Breathing Exercise on Anxiety and Pain in Patients Undergoing Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulku Gunes (Other)
Responsible Party: Sponsor-Investigator, Ulku Gunes, Profesor, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E10208771
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Procedural Pain; Procedural Anxiety
MeSH Terms: conditions — Pain, Procedural | interventions — Music Therapy; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: This single-center, single-blind, randomized controlled trial was conducted in Izmir, Turkey, from July 2021 to July 2022. Participants were randomly assigned to one of three groups: intervention 1 (music), intervention 2 (breathing exercises), or control (standard care), in a 1:1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: The nurse responsible for conducting all measurements, including pain and anxiety assessments using the Visual Analog Scale (VAS) and State-Trait Anxiety Inventory (STAI), was not part of the research team.
  The nurse, being independent and not aware of the participants' group assignments, helps to ensure that the assessments are conducted impartially, without knowledge of which intervention each participant received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music therapy (Active Comparator): After the patient was taken to the angiography laboratory, music was played using a digital MP3 player approximately 10 minutes before the angiography procedure began.
  Interventions: Behavioral: Music therapy
- Breathing exercise (Active Comparator): Individuals in the breathing exercise group were made to do breathing exercises by the researcher in the patient room 30 minutes before coronary angiography
  Interventions: Behavioral: Breathing exercise
- Control Group (No Intervention): All data collection steps were applied identically to the control group patients, except for music application and deep breathing exercises. All patients in the study group received the same routine care.

INTERVENTIONS:
Behavioral: Music therapy — After the patient was admitted to the angiography laboratory, approximately 10 minutes before the angiography procedure commenced, they were seated and allowed to relax. Music was played using a digital MP3 player.
  Arms: Music therapy
Behavioral: Breathing exercise — Individuals in the breathing exercise group were made to do breathing exercises by the researcher in the patient room 30 minutes before coronary angiography. The exercises were performed in a single patient room, in a quiet and calm environment. During the first 5 minutes, the researcher explained how the exercise was done with pictures and showed it to the patient. The patient was then asked to do the exercise for 10 minutes under the supervision of the researcher.
  Arms: Breathing exercise

SUMMARY:
Coronary angiography serves as the primary diagnostic technique for cardiovascular disease. However, this invasive procedure commonly triggers pain, anxiety, and fear in patients. The objective of this randomized controlled trial was to examine the impact of music and breathing exercises on anxiety and pain levels in individuals undergoing coronary angiography. The study, conducted as a single-blind, randomized controlled trial, involved a sample of 165 patients, with 55 in each group: the control group, the breathing exercise group, and the music therapy group. Patients in the music group listened to music during angiography, those in the breathing exercise group practiced exercises 30 minutes before the procedure, while the control group received standard treatment. Anxiety levels were assessed both before and after the procedure, and pain levels were measured post-procedure. The study strictly adhered to the CONSORT statement guidelines.

DETAILED DESCRIPTION:
Breathing exercises and music therapy have been demonstrated to be used in managing anxiety and pain in many clinical conditions, only a few studies have investigated their effectiveness on anxiety and pain during coronary angiography. Pain and anxiety are commonly experienced symptoms during coronary angiography. Therefore, the objective of this study is to examine the effects of the music and breathing exercises on anxiety and pain in patients undergoing coronary angiography.

Design This single-center, single-blind, randomized controlled trial was conducted in Izmir, Turkey, from July 2021 to July 2022. Participants were randomly assigned to one of three groups: intervention 1 (music), intervention 2 (breathing exercises), or control (standard care), in a 1:1:1 ratio. The study received approval from the Ethics Review Committee of a university hospital, and written informed consent was obtained from each participant.

Sample The participants were selected by the researcher from patients who were scheduled to undergo coronary angiography at the Cardiology clinic of a university hospital. Patients were included in the study if they met the following criteria: being scheduled for their first coronary angiography, being above 18 years of age, not being dependent on drugs or alcohol, having orientation to time and place, not experiencing respiratory distress, not having a history of serious psychological problems in the past 6 months, not taking any medication that suppresses anxiety symptoms and pain, and consenting to participate in the study. Patients who did not like music due to cultural reasons, stents implanted during angioplasty, required urgent treatment for the management of cardiac arrhythmias, had hearing problems, or had difficulty performing breathing exercises were excluded.

The sample size was calculated based on previous research on the effects of coronary angiography on pain and anxiety as well as our pilot study. We aimed to have a sufficient sample size to detect a difference of 2 units (mean ± SD) in pain levels between the intervention and control groups. 165 subjects were targeted for this study.

2.3. Randomization Eligible participants were randomly assigned to either the intervention groups or control group in a 1:1 ratio using a permuted block randomization method with a block size of 6. A random allocation sequence was generated by an off-site statistician who was not involved in participant recruitment. Allocation concealment was ensured by employing sealed opaque envelopes containing sequence numbers.

Intervention Breathing Group

Individuals in the breathing exercise group were made to do breathing exercises by the researcher in the patient room 30 minutes before coronary angiography. The exercises were performed in a single patient room, in a quiet and calm environment. During the first 5 minutes, the researcher explained how the exercise was done with pictures and showed it to the patient. The patient was then asked to do the exercise for 10 minutes under the supervision of the researcher. If the patient performed the Deep Breathing Exercise correctly, the application was terminated. If unable, the patient was asked to practice for another 5 minutes. If the patient still could not perform the exercise correctly after this period, he was excluded from the sample. Deep Breathing Exercise was applied according to the Cleveland Clinic Guideline. The Cleveland Clinic guide showed how to do the Deep Breathing Exercise with the knee bent. The following protocol was followed in the breathing exercise:

1. Ensure the patient is comfortably seated with bent knees, and relax the shoulders, head, and neck.
2. Place one hand on the upper chest and the other below the rib cage to enable the patient to sense diaphragm movement.
3. Initiate slow inhalation through the nose, allowing the abdominal region to expand outward.
4. Maintain stability in the hand on the chest to minimize movement.
5. Tighten the stomach muscles and exhale through pursed lips, facilitating the inward movement of the abdominal area.
6. Keep the hand on the upper chest as stable as possible throughout the process.

Music Group After the patient was admitted to the angiography laboratory, approximately 10 minutes before the angiography procedure commenced, they were seated and allowed to relax. Music was played using a digital MP3 player. The music was compiled from Johann Sebastian Bach's light instrumental music albums. Previous studies have demonstrated that this album has a positive impact on the cardiovascular system. The duration of music listening ranged from 20 to 40 minutes depending on the length of the procedure. Since the patient could be given coughing instructions during the procedure, headphones could not be used. Individuals lying on the bed in the angiography room were instructed to assume a comfortable position and focus on the music.

Control Group All data collection steps were applied identically to the control group patients, except for music application and deep breathing exercises. All patients in the study group received the same routine care.

Instruments Demographic variables and health characteristics of participants Demographic variables, such as age, education, marital status, and health characteristics (presence of chronic illnesses, coping mechanisms for stress, previous surgery history) were collected using a structured questionnaire.

State-Trait Anxiety Inventory State-Trait Anxiety Inventory (STAI), originally developed by Spielberg et al. to assess state and trait anxiety levels separately, has been adapted into the Turkish language by Öner and Le Compte. Validation and reliability studies for the Turkish version have been conducted, confirming its robustness. The scale consists of 40 items, with 20 items measuring state anxiety and 20 items measuring trait anxiety. Respondents were instructed to choose the response that best fits each item on the scale: "almost never," "sometimes," "often," or "almost always." Higher scores on the scale indicate greater levels of anxiety.

Visual Analog Scale It is a scale used to assess pain intensity. Visual Analog Scale (VAS) is stated to be more sensitive and reliable in measuring pain intensity compared to other single-dimensional scales. The VAS is a 10 cm ruler that can be used horizontally and vertically, with "0" representing no pain at one end and "10" representing the most severe pain at the other end. The patient marks the level of pain intensity they are experiencing on this ruler. Pain severity scores were measured in millimetres.

Outcome measures The primary outcome measurement is the patients' pain and anxiety levels. Individuals were assigned to the study groups after being informed about the research and obtaining their written consent. Initially, basic patient information was collected and recorded on the "Patient Identification Form". Subsequently, individuals were provided with information on the use of the VAS and the angiography procedure. Following this, individuals were assessed using the STAI. Afterwards, patients were taken to the angiography laboratory. Immediately after the angiography procedure was completed, the individuals' pain levels were evaluated and documented using the VAS. Thirty minutes after the angiography procedure was completed, individuals underwent an assessment using the STAI. All of these measurements were conducted by a nurse who was not part of the research team.

ELIGIBILITY:
Inclusion Criteria:

* being scheduled for their first coronary angiography
* being above 18 years of age
* not being dependent on drugs or alcohol
* having orientation to time and place
* not experiencing respiratory distress
* not having a history of serious psychological problems in the past 6 months
* not taking any medication that suppresses anxiety symptoms and pain

Exclusion Criteria:

* Patients who did not like music due to cultural reasons
* stents implanted during angioplasty
* required urgent treatment for the management of cardiac arrhythmias
* had hearing problems,
* had difficulty performing breathing exercises

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — It is based on self-representation of gender identity
Enrollment: 512 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | an average of 6 months
  State-Trait Anxiety Inventory (STAI), originally developed by Spielberg et al. to assess state and trait anxiety levels separately, has been adapted into the Turkish language by Öner and Le Compte. Validation and reliability studies for the Turkish version have been conducted, confirming its robustness. The scale consists of 40 items, with 20 items measuring state anxiety and 20 items measuring trait anxiety. Respondents were instructed to choose the response that best fits each item on the scale: "almost never," "sometimes," "often," or "almost always." Higher scores on the scale indicate greater levels of anxiety
Visual Analog Scale | an average of 6 months
  It is a scale used to assess pain intensity. Visual Analog Scale (VAS) is stated to be more sensitive and reliable in measuring pain intensity compared to other single-dimensional scales. The VAS is a 10 cm ruler that can be used horizontally and vertically, with "0" representing no pain at one end and "10" representing the most severe pain at the other end. The patient marks the level of pain intensity they are experiencing on this ruler. Pain severity scores were measured in millimetres.

CONTACTS AND LOCATIONS:
Overall Officials: ülkü güneş, Prof., Study Director — Ege University
Locations (2):
- Turkey (Türkiye) (2):
  - Ege University, Bornova, İzmir
  - Ülkü Güneş, Bornova, İzmir

REFERENCES:
- [Result] Oyur Celik G, Guzelcicek A, Celik S. The Effects of Music Therapy on Patients With Coronary Artery Disease Before the Invasive Procedure: A Randomized Controlled Study. J Perianesth Nurs. 2022 Apr;37(2):194-198. doi: 10.1016/j.jopan.2021.01.010. Epub 2021 Dec 28. PMID 34969619
- [Result] Ho CY, Wexberg P, Schneider B, Stollberger C. Effect of music on patients with cardiovascular diseases and during cardiovascular interventions : A systematic review. Wien Klin Wochenschr. 2021 Aug;133(15-16):790-801. doi: 10.1007/s00508-020-01782-y. Epub 2020 Dec 9. PMID 33296028
- [Result] Ebrahimi R, Shroyer AL, Dennis P, Currier J, Lendvai Wischik D. Music Can Reduce the Need for Pharmacologic Conscious Sedation During Invasive Coronary Angiography. J Invasive Cardiol. 2020 Nov;32(11):440-444. doi: 10.25270/jic/20.00132. Epub 2020 Oct 22. PMID 33087584
- [Result] Baljon KJ, Romli MH, Ismail AH, Khuan L, Chew BH. Effectiveness of breathing exercises, foot reflexology and back massage (BRM) on labour pain, anxiety, duration, satisfaction, stress hormones and newborn outcomes among primigravidae during the first stage of labour in Saudi Arabia: a study protocol for a randomised controlled trial. BMJ Open. 2020 Jun 15;10(6):e033844. doi: 10.1136/bmjopen-2019-033844. PMID 32540887
- See also: The Effects of Music Therapy on Patients With Coronary Artery Disease Before the Invasive Procedure: A Randomized Controlled Study — https://pubmed.ncbi.nlm.nih.gov/34969619/
- See also: Effect of music on patients with cardiovascular diseases and during cardiovascular interventions : A systematic review — https://pubmed.ncbi.nlm.nih.gov/33296028/
- See also: Music Can Reduce the Need for Pharmacologic Conscious Sedation During Invasive Coronary Angiography — https://pubmed.ncbi.nlm.nih.gov/33087584/
- See also: Effectiveness of breathing exercises, foot reflexology and back massage — https://pubmed.ncbi.nlm.nih.gov/32540887/